CLINICAL TRIAL: NCT05109936
Title: Non-inferiority Study of a New Therapeutic Strategy for Gout: Immediate Prescription of a Hypouricemic Treatment, Febuxostat, Compared to Its Delayed Administration - FEFACRIGOU Trial
Brief Title: Immediate Prescription of a Hypouricemic Treatment, Febuxostat, Compared to Its Delayed Administration
Acronym: FEFACRIGOU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/0386/HP
Record Dates: First submitted 2021-09-27; First posted 2021-11-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Immediate prescription (at randomization) of ADENURIC 80 mg / day (febuxostat), urate-lowering treatment, for a period of 2 x 6 weeks.
  Interventions: Drug: Adenuric
- Standard care arm (No Intervention): Prescription deferred to 6 weeks (42 days +/- 3 days) of ADENURIC 80 mg / day (febuxostat): hypouricemic treatment, for a period of 6 weeks.

INTERVENTIONS:
Drug: Adenuric — Immediate prescription (at randomization) of ADENURIC 80 mg / day (febuxostat), hypo-uricemic treatment, for a period of 2 x 6 weeks
  Arms: Experimental arm

SUMMARY:
Gout, the most common inflammatory rheumatism in France, is a complication of chronic hyperuricemia (> 360umol / l). The resulting urate crystals are deposited in many tissues, especially the skeletal or kidneys. It appears in the form of spontaneously regressive inflammatory joint attacks in 5 to 7 days but recurrent. Gout turns into a chronic disease if uric acidemia is not reduced, and is responsible for joint destruction. It becomes a vector of renal failure and is associated with cardiovascular morbidity and a reduction in life expectancy. It is cured if a long-term treatment such as febuxostat leading to the normalization of the uric acidemia is administered.

However, the frequency of this disease is increasing in industrialized or emerging countries. The causes are numerous, particularly food, but also related to flaws in therapeutic care. Studies show that this treatment is not taken in particular because, after the acute attack, the patient who has become asymptomatic again no longer consults. Currently, in a traditional way and according to European recommendations, it is not prescribed until several weeks after the acute attack in order to avoid early relapses, which would then be more numerous. Nevertheless, even if the hypouricemic agent is prescribed late , the attacks can be repeated and become rare for several months after obtaining a uricemia below 360umol / l; they eventually disappear. Lack of knowledge of this disease largely affects the hazards of disease-modifying treatment, which alone can prevent the progression to chronic inflammatory disease and its cardiovascular and renal impact and on mortality. One of the causes of not taking a hypouricemic agent is its delayed administration.

This study is proposed to assess the relevance of early initiation versus delayed administration of such treatment.

DETAILED DESCRIPTION:
This is a non-inferiority study comparing immediate administration with 6 weeks delayed administration of febuxostat at a dose of 80 mg / day. The methodology of non-inferiority is what we want to show. Indeed, the immediate initiation of a hypo-uricemic agent is currently considered as an aggravating factor with respect to the duration or the risks of early relapse of the crisis, without this being supported by precise studies. The basic treatment is beneficial in the long term: by normalizing uricemia, it controls gouty disease. We want to show that the early introduction is as well tolerated as its abstention which is the current recommendation.

The diagnosis of gout attack is based on recently established American-European criteria.

The choice of the hyporuricemic molecule is febuxostat, on the one hand because of a greater potency of action than allopurinol at the available dosages, which should make it possible to obtain a clear reduction in uraemia (of approximately 40%) and on the other hand easy to use - without dose adjustment - in patients with renal insufficiency with a creatinine clearance greater than 30 ml / min.

The number of patients participating in the study is set at 128, which is higher than the published prospective studies. Patients will be randomized (in order of succession when entering the study) into 2 groups, the first receiving febuxostat immediately for 6 weeks, the second receiving no immediate febuxostat treatment - which corresponds to current practice.

This study covers several periods:

* the first, lasting 6 weeks, will allow a direct comparison of febuxostat with no DMARD: this is the primary objective.
* the second is an extension phase and runs from the 7th to the 12th week where each patient in the context of routine care is treated with febuxostat: it makes it possible to compare the immediate use of the febuxostat (phase S0-S1 of the group 1) to its delayed administration (phase S6-S12 of group 2 with delayed administration) in terms of recurrence of gouty attacks.
* the 3 ° of 3 months allows a later evaluation at 6 months of therapeutic maintenance.

The evaluations will take place at the end of the 2nd and 6th week (plus or minus 3 days) and at the end of the 3rd and 6th month (plus or minus one week).

They are carried out by an assessor who does not know the treatment of the patient.

They are based on the following parameters:

1- The number of days with gouty joint crisis, its location, reported by the patient in a booklet filled out daily: the occurrence of a new attack according to the criteria evaluated will also be collected.

2 - Assessment by the patient of his condition (pain, asthenia, walking, overall condition) by daily use of the VAS scale. Two functional indexes will be used and have been evaluated in gout -: the SF 36 Physical Dimension is filled during the 6 ° and 12 ° week visits: this index was chosen because it was not specific for a joint disease. and evaluate a period of 4 weeks; HAQ, developed for rheumatoid arthritis, evaluates a period of 2 weeks and provides a correct estimate of overall physical function (locomotor status) in tophaceae gout, less in the absence of tophus.

3 - Assessment by the doctor of the patient's clinical condition: joint and somatic examination: arthritis (yes or no), presence of tophi, arterial pressure, cardiovascular and skin examination.

4 - Collection of drug intolerances. 5 - At W6 and W12, biological examinations will be carried out, according to the recommendations: determination of uricemia, serum creatinine, transaminases, CRP and determination of the CBC-platelets which makes it possible to control the intake and the biological tolerance of the hypouricemic treatment, the level of biological inflammation.

The treatment of the crisis will respond to European recommendations and will be left to the doctor's free initiative. This treatment will be immediately followed by a preventive treatment for relapse at the recommended doses.

Febuxostat:

Its indication will not refer to European recommendations but to French recommendations: hypo-uricemic treatment is indicated as soon as the diagnosis of gout is retained. It will be delivered at the same time as the treatment of the crisis, within 5 days maximum following its diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an attack of gout, diagnosed immediately or less than 5 days old. Gout is defined according to American-European criteria (Appendix 3).
2. Attack of gout affecting one (or more) peripheral joint (s) whatever (s) it (s):

   * Either a first crisis,
   * Either a new attack of a gout not treated with a hypo-uricemic or for which the hypo-uricemic treatment has not been taken for at least 6 months.
3. Uricemia ≥ 420 µmol / l, including under a diuretic (dosage carried out within 10 days before inclusion),
4. Age ≥ 18 years old,
5. Patient with a creatinine clearance ≥ 30 ml / min (dosage carried out within 10 days before inclusion),
6. Patient having read and understood the information letter and signed the consent form,
7. Affiliation to a social security scheme,
8. Woman of childbearing potential with effective contraception according to WHO definition (estrogen-progestins or intrauterine device or tubal ligation for more than 1 month and to be continued for at least 5 weeks after the last dose of the drug. ) and a negative urine pregnancy test on inclusion and throughout the duration of the study Where Postmenopausal woman: amenorrhea not medically induced for at least 12 months before the inclusion visit.

Exclusion Criteria:

1. Patients under the age of 18,
2. Stop taking a hypouricemic agent for less than 6 months,
3. Known contraindication to ADENURIC 80 mg film-coated tablet: hypersensitivity to the active substance (febuxostat) or to one of the excipients,
4. Renal failure defined by creatinine clearance <30 ml / min,
5. Hepatic disease defined by an increase to more than 2 times the normal of transaminases, alkaline phosphatases, to more than 3 times the normal of gamma-GT,
6. Non-weaned alcoholism,
7. Crisis more than 5 days old,
8. Patient who has received an organ or marrow transplant,
9. Person on Naproxen, mercaptopurine, azathioprine, Glycuronidation inhibitors and inducers, theophylline, macrolides, HMG Co-A reductase inhibitors and / or diuretic in combination with an ACE inhibitor or ARAII,
10. Person with rare hereditary disorders of galactose intolerance, lactase deficiency or glucose / galactose malabsorption
11. Poor understanding of the project due to neurological disease or lack of French practice,
12. Pregnant woman or likely to be in the absence of effective contraception (Women of childbearing age should have a negative urine pregnancy test),
13. Breastfeeding woman
14. Any history of pre-existing major cardiovascular disease (myocardial infarction, stroke, unstable angina, etc.), metabolic, endocrine, psychiatric or cancerous in uncontrolled development,
15. Person deprived of liberty by an administrative or judicial decision,
16. Person placed under judicial protection, guardianship or curatorship,
17. Participating patient who participated in the month preceding inclusion in another interventional drug trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the number of days with gout at 42 days +/- 3 days (W6) in patients with an early administration of febuxostat from the acute attack compared to patients with a delayed administration of febuxostat by 6 weeks after the acute attack. | 6 weeks
  number of days with gout at 42 days (S6) assessed by the daily booklet given to the patient, allowing him to inform daily whether he has suffered from gout or not

SECONDARY OUTCOMES:
To compare, in patients with early administration of febuxostat compared to patients with delayed administration the function of the patient during the study (until 26 weeks) | During the study (from the randomisation to 26 weeks)
  Physicians Global Assessment to measure quality of life
To compare, in patients with early administration of febuxostat compared to patients with delayed administration the intensity of pain during the study (until 26 weeks) | During the study (from the randomisation to 26 weeks)
  Visual Analog Score for pain
To compare, in patients with early administration of febuxostat compared to patients with delayed administration the tolerance of treatment during the study (until 26 weeks) | During the study (from the randomisation to 26 weeks)
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU de Caen, Caen
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - CHG Dieppe, Dieppe
  - CHI Elbeuf, Louvier, Val de Reuil, Elbeuf
  - GH Le Havre, Le Havre
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No